CLINICAL TRIAL: NCT02364154
Title: Metabolic Phenotyping of Blood Plasma by Means of 1H-NMR Spectroscopy: a New Tool to Detect Colorectal Cancer?
Brief Title: Colorectal Cancer Detected by 1H-NMR Spectroscopy
Acronym: BIOCOR
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Prof. dr. Michiel Thomeer, prof. dr., Hasselt University
Other Study IDs: 14/070U
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer
Keywords: biomarker; screening; coloscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples Without DNA — * blood plasma for NMR spectroscopy
  * blood sample for free circulating miRNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group-Blood sampling: -subjects with a normal colonoscopy
  Interventions: Other: Control group-Blood sampling; Other: Blood sampling
- Study group-Blood sampling: - subjects with colorectal cancer after colonoscopy
  Interventions: Other: Control group-Blood sampling; Other: Blood sampling

INTERVENTIONS:
Other: Control group-Blood sampling — Determine the metabolic phenotype of blood plasma by NMR spectroscopy
  Other Names: Metabolic phenotype
Other: Blood sampling — determine amount and type of free circulating miRNA in blood plasma
  Other Names: free circulating miRNA

SUMMARY:
The hypothesis of the present study is that metabolic phenotyping of blood plasma allows to (i) discriminate between colorectal cancer patients and control subjects and (ii) identify new biomarkers for colorectal cancer. In order to test this hypothesis, the investigators will apply proton nuclear magnetic resonance (1H-NMR) spectroscopy to perform metabolic phenotyping of blood plasma in 50 colorectal cancer patients and 50 control subjects. Multivariate statistics will be performed to assess the discriminative power of the applied methodology in distinguishing between both groups and to identify metabolites with potential as biomarkers for colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common and deadliest cancers worldwide. Since tumor stage at time of diagnosis is a critical determinant of patient outcome, early detection of colorectal cancer by screening modalities holds the key to improving patient survival. However, current tests, i.e. fecal occult blood testing and colonoscopy, are inadequate for first line screening of colorectal cancer due to limited accuracy and low participation rates, respectively. Therefore, there is an urgent need for new and accurate tests that can be used for en masse screening of colorectal cancer. A blood-based test represents a promising alternative as it takes little time, poses minimal risk to the patient, and is therefore very likely to lead to high participation rates. The development of an effective blood-based screening tool is based on the identification of biomarkers in the blood that are sensitive and specific for colorectal cancer. Studying the metabolic phenotype of colorectal cancer may help to identify such biomarkers since the metabolism of cancer cells is known to differ significantly from that of normal cells. More specifically, the entire metabolism of cancer cells is reprogrammed to increase anabolic reactions that favor cell growth and cell survival.

The hypothesis of the present study is that metabolic phenotyping of blood plasma allows to (i) discriminate between colorectal cancer patients and control subjects and (ii) identify new biomarkers for colorectal cancer. In order to test this hypothesis, The investigators will apply proton nuclear magnetic resonance (1H-NMR) spectroscopy to perform metabolic phenotyping of blood plasma in 50 colorectal cancer patients and 50 control subjects. Multivariate statistics will be performed to assess the discriminative power of the applied methodology in distinguishing between both groups and to identify metabolites with potential as biomarkers for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject has undergone a colonoscopy or is scheduled to undergo a colonoscopy in the future
* The subject is aged between 40 and 90 years
* The subject understands the study-specific procedures and provides written informed consent before any study-specific procedures are performed

Exclusion Criteria:

* No fasting starting from 10 p.m. the day prior to blood sampling
* Medication intake on the morning of blood sampling
* Diabetes
* History of cancer during the past 5 years
* Treatment for cancer during the past 5 years
* Inflammatory bowel disease

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients and control subjects who undergo a coloscopy without diabetes and/or a history of cancer during the past 5 years, of an age between 40 and 90 years and willing to provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
metabolic phenotype of colorectal cancer | day 1
  Significant metabolic changes in blood plasma of colorectal cancer patients compared with control subjects

SECONDARY OUTCOMES:
tumor histology | day 1
  subtype of histology of the colorectal tumor (according to WHO histological classification of tumors of the colon and rectum)
tumor stage | Day 1
  stage of the colorectal tumor, defined by the TNM classification system (7th edition)

CONTACTS AND LOCATIONS:
Overall Officials: Michiel thomeer, prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg, Hasselt University; Liesbet Mesotten, prof. dr., Study Chair — Ziekenhuis Oost-Limburg, Hasselt University; Philip Caenepeel, prof. dr., Study Chair — Ziekenhuis Oost-Limburg, Hasselt University; Peter Adriaensens, prof. dr., Study Chair — Hasselt University; Kirsten Stinkens, dr., Study Chair — Hasselt University; Evelyne Louis, PhD student, Study Chair — Hasselt University; Robby Louis, student, Study Chair — Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Background] Zhang A, Sun H, Yan G, Wang P, Han Y, Wang X. Metabolomics in diagnosis and biomarker discovery of colorectal cancer. Cancer Lett. 2014 Apr 1;345(1):17-20. doi: 10.1016/j.canlet.2013.11.011. Epub 2013 Dec 11. PMID 24333717
- [Background] Wang H, Wang L, Zhang H, Deng P, Chen J, Zhou B, Hu J, Zou J, Lu W, Xiang P, Wu T, Shao X, Li Y, Zhou Z, Zhao YL. (1)H NMR-based metabolic profiling of human rectal cancer tissue. Mol Cancer. 2013 Oct 18;12(1):121. doi: 10.1186/1476-4598-12-121. PMID 24138801
- [Background] Zavoral M, Suchanek S, Majek O, Fric P, Minarikova P, Minarik M, Seifert B, Dusek L. Colorectal cancer screening: 20 years of development and recent progress. World J Gastroenterol. 2014 Apr 14;20(14):3825-34. doi: 10.3748/wjg.v20.i14.3825. PMID 24744575
- [Background] Ganepola GA, Nizin J, Rutledge JR, Chang DH. Use of blood-based biomarkers for early diagnosis and surveillance of colorectal cancer. World J Gastrointest Oncol. 2014 Apr 15;6(4):83-97. doi: 10.4251/wjgo.v6.i4.83. PMID 24734154
- [Background] Beckonert O, Keun HC, Ebbels TM, Bundy J, Holmes E, Lindon JC, Nicholson JK. Metabolic profiling, metabolomic and metabonomic procedures for NMR spectroscopy of urine, plasma, serum and tissue extracts. Nat Protoc. 2007;2(11):2692-703. doi: 10.1038/nprot.2007.376. PMID 18007604
- [Result] Louis R, Louis E, Stinkens K, Mesotten L, de Jonge E, et al. (2016) Metabolic Phenotyping of Blood Plasma by Proton Nuclear Magnetic Resonance to Discriminate between Colorectal Cancer, Breast Cancer and Lung Cancer. Metabolomics (Los Angel) 6: 187. doi: 10.4172/2153-0769.1000187
- See also: Metabolic Phenotyping of Blood Plasma by Proton Nuclear Magnetic Resonance to Discriminate between Colorectal Cancer, Breast Cancer and Lung Cancer — https://www.omicsonline.org/open-access/metabolic-phenotyping-of-blood-plasma-by-proton-nuclear-magnetic-resonance-to-discriminate-between-colorectal-cancer-breast-cancer-2153-0769-1000187.pdf